CLINICAL TRIAL: NCT05260866
Title: Impact of the COVID-19 Pandemic on Mental Health Service Utilization in Children and Adolescents
Acronym: MENTALPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Nationale de Recherche (ANR) National Research Agency (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANR-21-COVR-0010-01
Record Dates: First submitted 2022-02-17; First posted 2022-03-02 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-02

CONDITIONS: Mental Disorder, Child
Keywords: pediatrics; COVID 19 pandemic; mental health; psychotropic drug
MeSH Terms: conditions — Neurodevelopmental Disorders; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: national population-based study — No intervention

SUMMARY:
Mental health consequences of the COVID-19 pandemic may be vast and may potentially overwhelm the mental health system in a long-lasting manner. Evaluating the effects of the COVID-19 pandemic on mental health in vulnerable groups such as children and adolescents has become an immediate priority. The aim of this study is to evaluate the impact of COVID-19 pandemic on use of mental health resources namely 1) prescriptions of psychotropic medications and 2) mental health-related outpatient visits, hospitalizations and emergency department visits in children and adolescents in France. Secondary aim is to evaluate the impact of the pandemic on episodes of fatal and non-fatal self-harm episodes in the same population. This will be a population-based cohort study using data from healthcare claims, administrative medical and outpatient drug dispensation databases in France between January 1, 2016 and June 1, 2021. Findings will inform on the risk of upcoming outbreaks of mental disorders that can result in significant morbidity and mortality and guide timely targeted actions to improve mental health outcomes and wellbeing in the youngest.

DETAILED DESCRIPTION:
Mental health consequences of the COVID-19 pandemic may be vast and may potentially overwhelm the mental health system in a long-lasting manner. Evaluating the effects of the COVID-19 pandemic on mental health in vulnerable groups such as children and adolescents has become an immediate priority. The aim of this study is to evaluate the impact of COVID-19 pandemic on use of mental health resources namely 1) prescriptions of psychotropic medications and 2) mental health-related outpatient visits, hospitalizations and emergency department visits in children and adolescents in France. Secondary aim is to evaluate the impact of the pandemic on episodes of fatal and non-fatal self-harm episodes in the same population. This will be a population-based cohort study using data from healthcare claims, administrative medical and outpatient drug dispensation databases in France between January 1, 2016 and June 1, 2021. Findings will inform on the risk of upcoming outbreaks of mental disorders that can result in significant morbidity and mortality and guide timely targeted actions to improve mental health outcomes and wellbeing in the youngest.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged from 6 to 18 years
* One dispensation of psychotropic medication or
* One mental-health related hospitalization or
* One reimbursement for an outpatient mental-health related consultation or
* One eligibility to long-term diseases corresponding to long term psychiatric diseases or
* One mental-health related cause of death using ICD-10 codes

Exclusion Criteria:

* none

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged from 6 to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of COVID-19 pandemic on use of mental health resources | 1 year
  prescriptions of psychotropic medications; mental health-related outpatient visits; mental health-related hospitalizations and emergency department visits

SECONDARY OUTCOMES:
To evaluate the impact of COVID-19 pandemic on episodes of fatal and non-fatal self-harm episodes in children and adolescents in France | 1 year
  monthly counts and rates of fatal and non-fatal self-harm episodes will be assessed throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Florentia Kaguelidou, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital - Assistance Publique Hopitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No